CLINICAL TRIAL: NCT00729417
Title: Obstetrical Risk Factors for the Development of Urinary and/or Fecal Incontinence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maaynei Hayesha Medical Center (Other)
Responsible Party: Obstetrical Risk Factors for the development of Urinary and/or Fecal Incontinence, Maaynei Hayeshua Medical Center
Other Study IDs: 0208
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Obstetric Risk Factors
Keywords: incontinence; obstetric risk factors; women; of age 18; above

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of Obstetrical Risk Factors for the development of Urinary and/or Fecal Incontinence according to a questionaire

The questionaire will be filled by the study investigators after the women participating in the study sign their consent. The study is based solely on a questionaire and does not include any physical examination, blood exam or intervention.

The study will be performed on the premises of Maaynei Hayeshua medical center. The inclusion criteria include women above the age of 18 who arrive to Maaynei Hayeshua Medical center for any reason. The data will be transferred to a computerized data base and analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* women of age 18 or above

Exclusion Criteria:

* women under the age of 18
* men

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women of age 18 or above
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-08 (Estimated)